CLINICAL TRIAL: NCT00949858
Title: New Data Analysis Methods for Actigraphy in Sleep Medicine
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Utah State University (Other)
Responsible Party: Sponsor
Other Study IDs: R01HL092347-01A1 (NIH)
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Obstructive Sleep Apnea; Restless Leg Syndrome; Insomnia
Keywords: Sleep Disorders; Obstructive Sleep Apnea; Restless Leg Syndrome; Insomnia; Actigraphy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Restless Legs Syndrome; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop statistical and informatics tools for analyzing and visualizing Actical™ (actigraphy) data linked to fatigue in Sleep Medicine Center patients.

DETAILED DESCRIPTION:
An Actical™ is a watch-like device attached to the wrist that uses an accelerometer to measure movement nearly continuously over several days. The American Academy of Sleep Medicine practice parameters report that actigraphy is a useful tool for detecting sleep in healthy individuals, assessing specific aspects in insomnia and restless legs syndrome, circadian-rhythm disorders, and excessive sleepiness. Concurrent with these recommendations is an increased interest in the use of actigraphy as a tool for objectively measuring fatigue. With improved high-end statistical methods for analyzing this data, actigraphy has the potential to become more important as an objective diagnostic tool for determining fatigue, sleep abnormalities and assessing response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting to the Washington University Sleep Medicine Center for evaluation of obstructive sleep apnea syndrome, restless legs syndrome, or insomnia
* Older than 18 years of age
* Ability to consent to participation in the study
* Willingness to wear the Actical™ for two 7 day periods and to return the equipment promptly

Exclusion Criteria:

* Inability to provide valid consent
* Pregnancy
* Night or rotating shift workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in clinic at the Washington University Sleep Medicine Center.
Sampling Method: Non-Probability Sample
Enrollment: 635 (Actual)
Dates: Start 2009-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01-22 (Actual)

PRIMARY OUTCOMES:
Define an object oriented data model for actigraphy and patient level data. | 6 months

SECONDARY OUTCOMES:
Apply existing and develop new advanced statistical and visualization methods for actigraphy data and include them in the data model listed above. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: William Shannon, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Sleep Medicine Center, St Louis, Missouri, United States